CLINICAL TRIAL: NCT01465971
Title: Monitoring of the Cerebral Tissue Oxygenation and Perfusion in the Adapting Climber During the Sleep in High Altitude
Brief Title: Monitoring of the Cerebral Tissue Oxygenation and Perfusion in the Adapting Climber During Sleep in High Altitude
Acronym: PerOxySleep
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Stein, Consultant of the Department for Anesthesiology, Intensive Care Medicine and Pain Therapy of the Goethe-University Frankfurt / Germany - Head of the working group for expedition medicine, Goethe University
Other Study IDs: ExpedMed#1-2011
Record Dates: First submitted 2011-10-26; First posted 2011-11-07 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Environmental Sleep Disorder; Cheyne-Stokes Respiration; Altitude Sickness
Keywords: high; altitude; acute; mountain; sickness; sleep; disorder; periodic; breathing; hyperventilation; apnea
MeSH Terms: conditions — Dyssomnias; Cheyne-Stokes Respiration; Altitude Sickness; Disease; Respiratory Aspiration; Hyperventilation; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- not acclimatized: no stay in an altitude above 2500 m within the last 3 Months
- acclimatized: stay above 2500 m with the last 14 days

SUMMARY:
One of the major challenges in adapting to high altitudes is that with increasing altitude sleeping quality declines rapidly. Thus, the night sleep can only provide limited to none regeneration. It usually takes a prolonged stay at a constant altitude to adapt sufficiently to the altitude and to have a refreshing night sleep. 1975 Reit et. al showed in their EEG-recordings that the sleep architecture (the regular succession of the particular sleep phases) is disturbed by repeating arousals which occur due to an irregularity in the breathing rhythm.

The purpose of this study is to create a better understanding of the underlying mechanisms that lead to failed acclimatization and AMS, due to sleep disturbance.

DETAILED DESCRIPTION:
Under sea level conditions humans breath between 10 and 12 times per minute. The breathing cycle in high altitude is accelerated. If the conscious breathing control vanishes during sleep a periodic breathing with alternating episodes of hyperventilation and apnea is the result. This circumstance causes repetitive arousals that do not allow a normal sleep pattern. The associated adverse effects are fatigue, slow or failed acclimatization, weakening of the immune system, lack of motivation and the disability to make rational decisions.

Sleep deprivation is a common reason for the abortion of a trip, accidents and severe forms of Acute Mountain Sickness (AMS).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 80 years
* voluntary participation in an expedition to Mount Kilimanjaro

Exclusion Criteria:

* obstructive or restrictive respiratory disorder
* hemodynamic relevant cardiac defect
* sleep disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants of an expedition to Mount Kilimanjaro
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation index | participants will be followed for the duration of the expedition, an expected 7 days
  Measured with near infra-red spectroscopy

SECONDARY OUTCOMES:
Tissue hemoglobin index | participants will be followed for the duration of the expedition, an expected 7 days
  measured with near infra-red spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stein, Dr.med., Principal Investigator — Goethe University
Locations (1):
- Clinic for Anaesthesia, Intensive Care Medicine and Pain Therapy, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Jackson SJ, Varley J, Sellers C, Josephs K, Codrington L, Duke G, Njelekela MA, Drummond G, Sutherland AI, Thompson AA, Baillie JK. Incidence and predictors of acute mountain sickness among trekkers on Mount Kilimanjaro. High Alt Med Biol. 2010 Fall;11(3):217-22. doi: 10.1089/ham.2010.1003. PMID 20919888
- [Background] Szymczak RK, Sitek EJ, Slawek JW, Basinski A, Sieminski M, Wieczorek D. Subjective sleep quality alterations at high altitude. Wilderness Environ Med. 2009 Winter;20(4):305-10. doi: 10.1580/1080-6032-020.004.0305. PMID 20030436
- See also: Working Group for Expeditionmedicine of the Goethe - University Frankfurt/Germany — http://www.expeditionsmedizin.de